CLINICAL TRIAL: NCT02587858
Title: NBIAready: Online Collection of Natural History Patient-reported Outcome Measures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Susan J. Hayflick (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor-Investigator, Susan J. Hayflick, Professor & Chair, Molecular & Medical Genetics, Oregon Health and Science University
Organization: Oregon Health and Science University (Other)
Other Study IDs: 10832
Record Dates: First submitted 2015-10-23; First posted 2015-10-27 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Neurodegeneration With Brain Iron Accumulation (NBIA)
Keywords: NBIA; PKAN; brain iron; Neurodegeneration with Brain Iron Accumulation; Hallervorden Spatz Syndrome; Pantothenate Kinase Associated Neurodegeneration; PLAN; INAD; PLA2G6-associated neurodegeneration; BPAN; Beta-propeller Protein-associated neurodegenration; WDR45; PLA2G6
MeSH Terms: conditions — Pantothenate Kinase-Associated Neurodegeneration; Neuroaxonal Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — BPAN participants will be asked for blood and saliva samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PKAN: This group consists of individuals diagnosed with PKAN using a combination of MRI, other clinical findings, and PANK2 gene sequencing.
- PLAN: This group consists of individuals diagnosed with PLAN using a combination of MRI, other clinical findings and PLA2G6 gene sequencing.
- BPAN: This group consists of individuals diagnosed with BPAN using a combinatino of MRI, other clinical findings, and WDR45 gene sequencing.

SUMMARY:
The purpose of this study is to learn more about Neurodegeneration with Brain Iron Accumulation (NBIA) Disorders. Data is being collected on three types of NBIA disorders:

Pantothenate Kinase-Associated Neurodegeneration (PKAN), PLA2G6-associated Neurodegeneration (PLAN) and Beta-propeller Protein-associated Neurodegeneration (BPAN). The study will (1) collect information about how symptoms and findings in NBIA change over time and (2) identify measures of NBIA that can be used in future clinical trials. Participants will follow links to a secure website every 6 months for a period of 5-10 years to electronically complete a set of rating scales as related to their NBIA disorder.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PKAN, PLAN or BPAN confirmed by gene testing and/or clinical features.
* Ability to access a computer with internet services or a phone approximately once every 6 months for up to 10 years to enter data.

Exclusion Criteria:

* Individuals who are not fluent in reading and communicating in English.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The PKAN group consists of international individuals diagnosed with PKAN. The PLAN group consists of international individuals diagnosed with PLAN. The BPAN group consists of international individuals diagnosed with BPAN.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-04; Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Document the natural history of NBIA and identify new markers of disease progression. | 5-10 years
  The unit of analyses will be the data collected on NBIA milestones and patient-reported outcome measures. Latent Growth Curve (LGC) modeling will be used to characterize the natural history of NBIA. If data support that certain disease milestones occur in a consistent order, or at consistent ages, then these data points will be candidate markers of disease progression. LGC will be used to characterize the natural history of NBIA and identify areas in which individuals with NBIA differ from the general population.

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Hayflick, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Official website of the OHSU NBIA research group — http://www.nbiacure.org